CLINICAL TRIAL: NCT03011528
Title: CombinaiR3 - First-line Treatment of Ewing Tumours With Primary Extrapulmonary Dissemination in Patients From 2 to 50 Years
Brief Title: First-line Treatment of Ewing Tumours With Primary Extrapulmonary Dissemination in Patients From 2 to 50 Years (CombinaiR3)
Acronym: CombinaiR3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IC 2015-13
Record Dates: First submitted 2016-12-06; First posted 2017-01-05 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Ewing Sarcoma Family of Tumors
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — Consolidation Chemotherapy; Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- VDC - IE x2 & Surgery (Other): Patients in Arm A receive
  * VDC-IE x2: Intensified induction phase:
    * 4 cycles of VDC (Vincristine Doxorubicine Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association if "good response" after the 4th treatment, followed by:
    * 4 cycles of VDC (Vincristine-Doxorubicine-Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association
  * Consolidation BuMel High dose chemotherapy (Busulfan Melphalan) followed by Peripheral Blood Stem Cell Infusion
  * Local treatment by surgery of primary tumour/metastatic sites (outside pulmonary sites): indicated before of after consolidation phase (BuMel) among multidisciplinary decision. Radiotherapy can be added
  * Maintenance phase
    * 1st year : VC (Vincristine Cyclophosphamide) association
    * 2nd year : Cyclophosphamide po 25 mg/m²
  Interventions: Drug: VDC-IE x2; Drug: Consolidation BuMel; Drug: Maintenance; Procedure: Local treatment by surgery; Radiation: Local treatment by radiotherapy
- VDC - IE & TEMIRI & Surgery (Other): Patients in Arm B receive
  * VDC-IE & TEMIRI: Intensified induction phase:
    * 4 cycles of VDC (Vincristine-Doxorubicine-Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association if "poor response" after the 4th treatment, followed by:
    * 4 cycles of TEMIRI (Temozolomide-Irinotecan) association
  * Local treatment by surgery of primary tumour/metastatic sites (outside pulmonary sites): indicated before of after consolidation phase (BuMel) among multidisciplinary decision. Radiotherapy can be added
  * Consolidation BuMel High dose chemotherapy (Busulfan-Melphalan) followed by Peripheral Blood Stem Cell Infusion
  * Maintenance phase
    * 1st year : VC (Vincristine Cyclophosphamide) association
    * 2nd year : Cyclophosphamide po 25 mg/m²
  Interventions: Drug: VDC-IE; Drug: TEMIRI; Drug: Consolidation BuMel; Drug: Maintenance; Procedure: Local treatment by surgery; Radiation: Local treatment by radiotherapy
- VDC - IE x2 & Radiotherapy (Other): Patients in Arm C receive
  * VDC-IE x2: Intensified induction phase:
    * 4 cycles of VDC (Vincristine-Doxorubicine-Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association if "good response" after the 4th treatment, followed by:
    * 4 cycles of VDC (Vincristine-Doxorubicine-Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association
  * Consolidation BuMel High dose chemotherapy (Busulfan-Melphalan) followed by Peripheral Blood Stem Cell Infusion
  * Local treatment by radiotherapy of primary tumour/metastatic sites (outside pulmonary sites): indicated before of after consolidation phase (BuMel) among multidisciplinary decision.
  * Consolidation BuMel High dose chemotherapy (Busulfan-Melphalan) followed by Peripheral Blood Stem Cell Infusion
  * Maintenance phase
    * 1st year : VC (Vincristine Cyclophosphamide) association
    * 2nd year : Cyclophosphamide po 25 mg/m²
  Interventions: Drug: VDC-IE x2; Drug: Consolidation BuMel; Drug: Maintenance; Radiation: Local treatment by radiotherapy
- VDC - IE & TEMIRI & Radiotherapy (Other): Patients in Arm D receive
  * VDC-IE & TEMIRI: Intensified induction phase:
    * 4 cycles of VDC (Vincristine-Doxorubicine-Cyclophosphamide) association alternative with 4 cycles of IE (Ifosfamide-Etoposide) association if "poor response" after the 4th treatment, followed by:
    * 4 cycles of TEMIRI (Temozolomide-Irinotecan) association
  * Local treatment by radiotherapy of primary tumour/metastatic sites (outside pulmonary sites): indicated before of after consolidation phase (BuMel) among multidisciplinary decision.
  * Consolidation BuMel High dose chemotherapy (Busulfan-Melphalan) followed by Peripheral Blood Stem Cell Infusion
  * Maintenance phase
    * 1st year : VC (Vincristine Cyclophosphamide) association
    * 2nd year : Cyclophosphamide po 25 mg/m²
  Interventions: Drug: VDC-IE; Drug: TEMIRI; Drug: Consolidation BuMel; Drug: Maintenance; Radiation: Local treatment by radiotherapy

INTERVENTIONS:
Drug: VDC-IE x2 — Week 1, 5, 9 and week 13:
  * Vincristine, IV, D1, 1.5mg/m²
  * Doxorubicine, IV, D1-D2, 37.5mg/m²
  * Cyclophosphamide, IV, D1, 1.2g/m²
  Week 3, 7, 11 and week 15:
  * Ifosfamide, IV, D15 to D19, 1.8g/m²/d
  * Etoposide, IV, D15 to D19, 100mg/m²/d
  Other Names: Intensified Induction VDC-IE x2
  Arms: VDC - IE x2 & Radiotherapy; VDC - IE x2 & Surgery
Drug: VDC-IE — Week 1 and week 5:
  * Vincristine, IV, D1, 1.5mg/m²
  * Doxorubicine, IV, D1-D2, 37.5mg/m²
  * Cyclophosphamide, IV, D1, 1.2g/m²
  Week 3, and week 7:
  * Ifosfamide, IV, D15 to D19, 1.8g/m²/d
  * Etoposide, IV, D15 to D19, 100mg/m²/d
  Other Names: Intensified Induction VDC-IE
  Arms: VDC - IE & TEMIRI & Radiotherapy; VDC - IE & TEMIRI & Surgery
Drug: TEMIRI — Week 9, 12, 15 and week 18:
  * Temozolomide, PO, D1 to D5, 150mg/m²/d
  * Irinotecan, IV, D1 to D5, 50mg/m²/d
  Other Names: Intensified Induction TEMIRI
  Arms: VDC - IE & TEMIRI & Radiotherapy; VDC - IE & TEMIRI & Surgery
Drug: Consolidation BuMel — After induction phase and local treatment (surgery and/or radiotherapy) and before PBSC:
  * Busulfan, IV, D-5 to D-2, dosa according to the weight
  * Melphalan, IV, D-1, 140 mg/m²
  Peripheral Blood Stem Cell infusion:
  - PBSC infusion, D0, at least 3.10^6 CD34/kg
  Other Names: High dose Consolidation chemotherapy
Drug: Maintenance — * 1st year : VC
  * Vinblastine, IV, 3mg/m², once a week (except during radiotherapy: 1mg/m², 3 times a week)
  * Cyclophosphamide, PO, 25mg/m² continuously
  Other Names: 2 years maintenance
Procedure: Local treatment by surgery — Surgical excision of whole site of the primary tumour and metastatic sites (outside pulmonary sites) can take place before or after the high dose consolidation chemotherapy. Radiotherapy can be added
  Other Names: Surgery of primary tumour/metastatic sites
  Arms: VDC - IE & TEMIRI & Surgery; VDC - IE x2 & Surgery
Radiation: Local treatment by radiotherapy — Radiotherapy of whole site of the primary tumour and metastatic sites (outside pulmonary sites) can take place before or after the high dose consolidation chemotherapy
  Other Names: Radiotherapy of primary tumour/metastatic sites

SUMMARY:
Ewing's sarcoma and related tumours (ESFT) are rare tumours, with a peak incidence in the second decade of life. They start most often from bone, and are characterized by a specific translocation involving the so-called EWS gene. In one patient out of three, the staging procedures detect metastatic tumours at the diagnosis, most commonly in lungs, bones, and bone marrow.

ESFT treatment strategy is multidisciplinary, combining primary chemotherapy, a local treatment, and consolidation chemotherapy.

The primary metastatic dissemination is the most important prognostic factor, as the survival rate is around 70-75% for localized tumours, in contrast with less than 50% for patients with primary metastatic disease.

Among primary metastatic patients, bone involvement and / or bone marrow strike markedly the prognosis of these patients. While the long-term survival of patients with isolated pleural pulmonary metastases is approximately 50%, whereas it is only from 0 to 25% in patients with bone marrow involvement.

In 1999, the Intergroup EURO EWING built a new study protocol for patients with Ewing tumours. For the patients with primary extrapulmonary metastatic Ewing tumours (R3 patients), the protocol proposed a heavy induction chemotherapy, in order to propose a consolidation with high dose chemotherapy to a higher rate of patients. The high-dose Busulfan Melphalan chemotherapy (BuMel) was based on Busulfan (600 mg/m²) and Melphalan (140 mg/m²), with autologous peripheral blood stem cell (PBSC) support.

Of note, for the full population of patients with metastatic disease, the 3-year EFS rate was 27% (SD 3%), and the OS rate was 34% (SD 4%), with a median follow-up of 3.9 years after diagnosis, and a median survival time of 1.6 years.

DETAILED DESCRIPTION:
Ewing's sarcoma and related tumours (ESFT) are rare tumours, with a peak incidence in the second decade of life. They start most often from bone, and are characterized by a specific translocation involving the so-called EWS gene. The gene rearrangement results in the production of a transcription factor, in the majority EWS-FLI1 transcription.

In one patient out of three, the staging procedures detect metastatic tumours at the diagnosis; metastases involve most commonly lungs, bones, and bone marrow.

Therefore, in addition to local imaging, the initial extension assessment of any Ewing tumour includes at least a chest CT scan, and a bone marrow extensive evaluation, comprising bone marrow punctures into several different sectors, bone marrow biopsies, and a bone imaging evaluation. The FDG-PET scan is more sensible than bone scan and conventional imaging as MRI in detection of bone metastases. It is more and more widely used in the bone metastasis search in Ewing tumours and seems useful to complement the search of extra-osseous metastases (outside the lungs), including that of bone marrow metastases. The full-body MRI is still under evaluation for the disease extension evaluation.

ESFT treatment strategy is multidisciplinary, combining primary chemotherapy, a local treatment, and consolidation chemotherapy. The local treatment may combine surgery and / or radiotherapy, according to the tumour site and size, and to the tumour response. ESFT chemotherapy is based on alkylating agents (ifosfamide and / or cyclophosphamide), etoposide, anthracyclines, vincristine, and actinomycin.

The primary metastatic dissemination is the most important prognostic factor, as the survival rate is around 70-75% for localized tumours, in contrast with less than 50% for patients with primary metastatic disease. Among primary metastatic patients, bone involvement and / or bone marrow strike markedly the prognosis of these patients. While the long-term survival of patients with isolated pleural pulmonary metastases is approximately 50%, whereas it is only from 0 to 25% in patients with bone marrow involvement.

In 1999, the Intergroup EURO EWING built a new study protocol for patients with Ewing tumours, localized or metastatic and below 50 years of age. For the patients with primary extrapulmonary metastatic Ewing tumours (R3 patients), the protocol proposed a heavy induction chemotherapy, in order to propose a consolidation with high dose chemotherapy to a higher rate of patients. The high-dose BuMel chemotherapy was based on Busulfan (600 mg/m²) and Melphalan (140 mg/m²), with autologous peripheral blood stem cell (PBSC) support.

The study enrolled 281 patients with primary dissemination and skeletal metastases, with or without bone marrow involvement and with or without additional pulmonary metastases or metastases to other sites. In contrast to the distribution in the entire group of patients with Ewing tumours, the primary site in this subgroup was extremity in only 31% patients, pelvis/abdomen in 45%, and axial/other in 24% patients. The overall survival at 3 years was 28% (SD 4%) in the group with primary tumour in the abdomen or pelvis, versus 39% (SD 6%) for each of the two other groups. Of note, for the full population of patients with metastatic disease, the 3-year EFS rate was 27% (SD 3%), and the OS rate was 34% (SD 4%), with a median follow-up of 3.9 years after diagnosis, and a median survival time of 1.6 years.

ELIGIBILITY:
Inclusion Criteria:

1. - Ewing tumour histologically or cytologically confirmed, harboring a specific transcript, and with extrapulmonary metastases (including nodal extension) - histology and FISH results must be consistent, specific transcript can be obtained after inclusions.
2. - Ewing tumour not previously treated.
3. - Age between 2 and 50 years.
4. - Measurable disease by cross sectional imaging (RECIST 1.1) or evaluable disease with functional metabolic, positron emission tomography scanner (PET SCAN) or other methods (e.g., cytology/histology).
5. - General status compatible with the study treatments (LANSKY score ≥ 50%, or Karnofsky ≥ 50%, or Eastern Cooperative Oncology Group (ECOG) ≤ 2).
6. - Adequate bone marrow function (not applicable in case of bone marrow disease).

   * Platelets ≥ 100 x 109 /L
   * Absolute Neutrophil Count (ANC) ≥ 1 x 109 /L
   * Hemoglobin ≥ 8g /dL.
7. - Adequate liver function :

   * Aspartate Aminotransferase (AST) and Alanine Transferase (ALT) ≤ 5 x Upper Limit Normal (ULN)
   * Total Bilirubin ≤ 2 Upper Limit Normal (ULN). If total bilirubin > 2xULN, Bilirubin Conjugated Fraction (BCF) ≤ 2 x ULN
8. - No absolute contra-indication of Busulfan-Melphalan if radiotherapy of the primary tumour is necessary with specific attention to patient with primary spinal tumor.
9. - Adequate cardiac and renal functions:

   * Creatinine < 1.5 of normal for age or clearance > 60 ml/min/1.73 m²;
   * Left Ventricular Ejection Fraction (LVEF) > 50% and/or shortening fraction > 28%.
10. - No underlying disease contra-indicating the study treatments.
11. - Patient likely compliant with the recommended study medical monitoring during and after treatments.
12. - Patients of childbearing potential must agree to use adequate contraception for the duration of study treatments and up to 12 months for women and 6 months for men following completion of therapy.
13. - Females of childbearing potential must have a negative serum β-human chorionic gonadotropin (HCG) pregnancy test within 10 days prior study inclusion, and/or urine pregnancy test within 48 hours before the first administration of the study treatment.
14. - Patients covered by a health insurance system.
15. - Patient, or patient's legal representative, informed and having signed the informed consent.

Exclusion Criteria:

1. - Age below 2 or greater than 50 years.
2. - Ewing tumour localized, or solely with pleural and/or lung metastases.
3. - Concomitant disease, particularly infectious disease, likely to interfere with patient's treatment.
4. - History of cancer, according to investigator's judgment.
5. - Life expectancy < 2 months.
6. - Patient already included in another clinical trial with an investigational drug.
7. - Pregnant or breastfeeding patient.
8. - Person deprived of liberty or under guardianship.
9. - Patient likely unable to comply with the study medical monitoring for geographical, social or psychological reasons.

Ages: 2 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-08 (Actual); Study Completion 2023-11 (Actual)

PRIMARY OUTCOMES:
Anti-tumour effect of the treatment strategy assessed by the number of patients event-free survival (EFS) at 18 months | 18 months after inclusion of the last patient
  EFS is defined as the time from inclusion date to the first documentation of progression, distant disease, second cancer or death (or last news for patients free of event). The event free survival is estimated by Kaplan-Meier method.

SECONDARY OUTCOMES:
Anti-tumour effect of the dose-intensified induction chemotherapy assessed by the response rate of patients | week 19-20 = Response Evaluation 2 (RE2)
  Number of patients with complete response (CR) / partial response (PR) eligible for consolidation phase
Anti-tumour effect of the dose-intensified induction chemotherapy assessed by the number of patients eligible for consolidation phase | week 19-20 = RE2
  Number of patients eligible for consolidation phase have good response after induction phase :
  * complete remission on primary tumour and on metastatic sites or
  * very good disease response defined by:
    * complete or partial response according to RECIST 1.1 criteria on primary lesion
    * complete or very good partial response (> 90 %) in case of RECIST 1.1 criteria on metastatic sites AND
    * complete metabolic response in case of metastatic visceral and/or bone/bone marrow lesions, or very good partial response according to investigator's judgment AND
    * in case of bone marrow involvement, bone marrow free of disease on at least one biopsy and two punctures at different sites at RE1 (evaluation after 4 cycles VDC-IE), RE2 (evaluation after 2x4 cycles VDC-IE or 4 cycles VDC-IE+4 cycles TEMIRI), or at the latest RE3 evaluation (evaluation after local treatment).
Overall survival (OS) is assessed by the number of patients still alive at the end of the three years of treatment | 3 years = Response Evaluation End-Of-Treatment (EOT RE)
  The overall survival (OS) is estimated by Kaplan-Meier method.
3-years event-free survival (EFS) is assessed by the number of patients without any event at the end of treatment phase | 3 years = EOT RE
  EFS is defined as the time from inclusion date to the first documentation of progression, distant disease, second cancer or death (or last news for patients free of event). The event free survival is estimated by Kaplan-Meier method.
Number of patients with treatment-related adverse events as assessed by CTCAE v4.03 | week 19-20 = RE2 ; week 27-28 = Response Evaluation 3 (RE3); 3 years = EOT RE
  Number of patients with treatment-related adverse events using the NCI CTCAE version 4.03 to graduate the severity of adverse events
Number of patients with treatment-related toxicities on laboratory data as assessed by CTCAE v4.03 of the different phases of treatment | week 19-20 = RE2 ; week 27-28 = RE3; 3 years = EOT RE
  Number of patients with treatment-related toxicities on laboratory data using the NCI CTCAE version 4.03 to graduate the severity of toxicities
18F-FDG PET evaluation efficacy assessed by primary tumour uptake | study inclusion, after week 8 (RE1), after week18-19 (if VDC-IE) or week19-20 (if TEMIRI)=RE2, after local treatment ≤week30 (RE3), from week31 (=RE4), 3 years = EOT RE
  Efficacy assessed by primary tumour uptake (Standardized Uptake Value max at 18F-FDG PET)
18F-FDG PET evaluation efficacy assessed by metabolic tumour volume (MTV) | study inclusion, after week 8 (RE1), after week18-19 (if VDC-IE) or week19-20 (if TEMIRI)=RE2, after local treatment ≤week30 (RE3), from week31 (=RE4), 3 years = EOT RE
  Efficacy assessed by metabolic tumour volume (MTV at 18F-FDG PET)
Percentage of circulating tumour cells in blood and bone marrow to correlate with patient outcome (EFS). Ancillary study | study inclusion, and/or during Procedure=surgery (if done) either after week 19-20=RE2 or after PBSC infusion=RE4
  sample collected : primary tumour and metastatic site (if possible)
Percentage of circulating tumour cells in blood and bone marrow to correlate with patient outcome (EFS). Ancillary study | study inclusion, at each evaluation time (RE1=week8 to Response Evaluation before maintenance therapy (RE5=<week38)), every 3 months during 2 years maintenance therapy, at End of Treatment
  sample collected : blood
Percentage of circulating tumour cells in blood and bone marrow to correlate with patient outcome (EFS). Ancillary study | at diagnosis (before treatment), at 1st evaluation time (RE1=wk8 if bone marrow involvement at diagnosis), at RE2=week19-20 (or RE3=<week30), after PBSC infusion=RE4 or RE5=< week38 (if bone marrow involvement at diagnosis), at End of Treatment
  sample collected : bone marrow
Comparison of transcriptomic profiles between those of primary disease and those of bone marrow metastases to determine if they are the same or not. Ancillary study | study inclusion
  Investigation whether the cells from metastatic material harbour a unique transcriptomic signature compared to primary tumour cells : quantification of EWS-ETS transcript and EWS-ETS gene using Polymerase Chain Reaction (PCR) methods to determine the genomic EWS-ETS translocation loci

CONTACTS AND LOCATIONS:
Overall Officials: Valérie LAURENCE, MD, Principal Investigator — Institut Curie; Nadège CORRADINI, MD, Principal Investigator — Institut d'Hématologie et d'Oncologie Pédiatrique
Locations (17):
- France (17):
  - Chr Felix Guyon, La Réunion, Saint Denis
  - Bordeaux Chu, Bordeaux
  - CHU Grenoble Alpes, Grenoble
  - LILLE Centre Oscar Lambret, Lille
  - LYON Centre Léon Bérard, Lyon
  - Marseille Chu, Marseille
  - CHRU Montpellier - Hôpital A. de Villeneuve, Montpellier
  - Nantes Chu, Nantes
  - PARIS Institut Curie, Paris
  - PARIS Trousseau, Paris
  - CHU Hôpital Sud, Rennes
  - Strasbourg Chu, Strasbourg
  - Toulouse Chu, Toulouse
  - TOULOUSE Institut Claudius Regaud, Toulouse
  - Nancy Chu, Vandœuvre-lès-Nancy
  - NANCY Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - VILLEJUIF Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).

REFERENCES:
- [Result] Laurence V, Jehanno N, Dureau S, Mous L, Claude L, Ballet S, Pierron G, Gaspar N, Brahmi M, Valentin T, Revon-Riviere G, Lervat C, Probert J, Entz-Werle N, Mansuy L, Plantaz D, Rios M, Saumet L, Verite C, Castex MP, Thebaud E, Cassou-Mounat T, Plissonnier AS, Dieppedale J, Delattre O, Legrier ME, Marec-Berard P, Gouin F, Berlanga P, Cordero C, Surdez D, Corradini N. Interest of a sequential multimodal approach for the treatment of newly diagnosed patients with multimetastatic Ewing sarcoma: results of the French prospective CombinaiR3 phase II trial. Br J Cancer. 2025 Nov 17. doi: 10.1038/s41416-025-03263-3. Online ahead of print. PMID 41249450